CLINICAL TRIAL: NCT04949867
Title: Dual-Hormone Closed-Loop Glucose Control in Adolescents With Type 1 Diabetes
Acronym: DHCL2021
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-21000207; 2020-005836-31 (EudraCT Number); 2021-0409-34 (Other: Eudramed CIV-ID-nr.); PD002-19 (Other Grant/Funding Number: Danish Diabetes Academy)
Record Dates: First submitted 2021-05-18; First posted 2021-07-02 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded, cross-over study of glycemic control during dual-hormone therapy compared with single-hormone therapy in adolescents with type 1 diabetes.
Who Masked: Participant
Masking Description: . For dual-hormone control, the study pumps will be filled with FiAsp® and GlucaGen®. For single-hormone control, the study pumps have been filled with FiAsp® and isotonic saline. Pump filling is conducted before the participant arrives at the research facility. The glucagon/saline pump and the insulin pump are clearly marked and cannot be confused. The participants are blinded to the treatment, as isotonic saline by its looks is indistinguishable from GlucaGen®. The placebo pump ('dummy' pump) will not infuse the saline and cannot be detected by the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-hormone Closed-loop (Active Comparator): FiAsp® and GlucaGen®.
  Interventions: Drug: Glucagon; Device: Closed-loop System
- Single-Hormone Closed-loop (Placebo Comparator): FiAsp® and isotonic saline.
  Interventions: Device: Closed-loop System

INTERVENTIONS:
Drug: Glucagon — Glucagon is filled in the pump and given automatically in case of hypoglycemia or pending hypoglycemia.
  Other Names: GlucaGen, Novo Nordisk,
  Arms: Dual-hormone Closed-loop
Device: Closed-loop System — Closed-loop system comprise of two DANA RS (R) insulin pumps (FiAsp-GlucaGen vs FiAsp-saline), one DexCom G6 sensor, and a smartphone for the control algorithm.
  Other Names: Saline

SUMMARY:
Objective:

To assess the efficacy and safety of an insulin-glucagon dual-hormone (DH) closed-loop system compared with an insulin-only single-hormone (SH) closed-loop system in adolescent with type 1 diabetes.

Methods:

In a 26-h, randomized, crossover, inpatient study, 20 children and adolescents with type 1 diabetes used two modes of the DiaCon Artificial Pancreas system: DH and SH closed-loop control. During each study period, participants will have one overnight stay, received three meals and performed exercise for 45 min (bicycle with estimated 50% V02max).

Endpoint:

The primary endpoint is sensor-derived percentage of time in hypoglycemia (<3.9 mmol/L).

DETAILED DESCRIPTION:
Upon arrival at the research facility at Steno Diabetes Center Copenhagen, the participant's own pump and CGM are disconnected, and the two study pumps are attached. For dual-hormone control, the study pumps will be filled with FiAsp® and GlucaGen®. For single-hormone control, the study pumps have been filled with FiAsp® and isotonic saline.

In addition, participants are provided with a blinded wearable activity and sleep monitoring device (ActiGraph GT9X Link, Pensacola, FL) for activity level estimation and sleep assessment during study participation. The Actigraph is connected to a Bluetooth® Polar heart rate monitors during the exercise session.

Female participants deliver a urine sample for pregnancy testing. A sampling cannula is placed in an antecubital vein. The CGM will be calibrated with fingerpick glucose meter (Contour next®, Ascensia Diabetes Care) before initiating the closed-loop control. Even though it is not needed to calibrate the sensor, the accuracy of the sensor is better after one calibration.

At day 1 17:00 the study is initiated, and the closed-loop system takes over glucose control. Except from the control approach (single- vs. dual-hormone), the study days are identical. During the study visit, participants can move around freely, but they can only perform actual exercise during the stationary bike exercise session at day 2 16:30. At nighttime, the participants are encouraged to be in bed and, if possible, sleep.

At predefined timepoints, the investigators measure blood pressure and pulse, and the investigators ask the participants to rate their nausea level on a visual analog scale (VAS) from 1 to 100 to assess possible side effects of glucagon (vomiting rates as 100). In addition, the investigators ask them to self-rate blood glucose levels before bedtime (23:00), upon wake-up (07:00-08:00), before each meal, before exercise, and every 10 minutes during exercise.

Single-hormone and dual-hormone closed-loop control study sessions end 26 hours after study start. The study pumps and the CGMs are disconnected and the participants reconnect their own pumps and CGMs.

The two study sessions are separated by at least 36 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age = 13-17 years
* T1D duration ≥ 2 years
* Insulin pump therapy ≥ 1 year
* Using CGM or isCGM (Flash Libre)
* HbA1c ≤ 9.0% (75 mmol/mol)
* Using carbohydrate counting

Exclusion Criteria:

* Allergy to glucagon or lactose
* Allergy to faster insulin aspart (FiAsp)
* Pheochromocytoma
* Self-reported lack of hypoglycemia symptoms when blood glucose is < 3.0 mmol/l
* Inability to follow study procedures, e.g. exercise, sleeping, blood sampling, and meal intake
* Pregnancy, nursing, plan to become pregnant or sexually active and not using adequate contraceptive methods (intrauterine device, contraceptive pill, patch or injection)
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during or within 30 days prior to study participation
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the participant unsuitable for study participation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage of time with glucose values < 3.9 mmol/l as measured by the continuous glucose monitor | 26 hours during closed-loop control
  Percentage

SECONDARY OUTCOMES:
Number of carbohydrate interventions to treat hypoglycemia | 26 hours during closed-loop control
Percentage of time with glucose values in the range 3.9-10.0 mmol/l measured by continuous glucose monitor and plasma glucose | 26 hours during closed-loop control
  Percentage
Percentage of time with glucose values < 3.9 mmol/l as measured by plasma glucose | 26 hours during closed-loop control
  Percentage
Percentage of time with glucose values in the range > 13.9 mmol/l measured by continuous glucose monitor and plasma glucose | 26 hours during closed-loop control
  Percentage
Percentage of time with glucose values < 3.0 mmol/l as measured by continuous glucose monitor and plasma glucose | 26 hours during closed-loop control
  Percentage
Mean blood glucose value measured by continuous glucose monitor and plasma glucose | 26 hours during closed-loop control
  mmol/L
Number of hypoglycemic episodes < 3.9 mmol/l on continuous glucose monitor and plasma glucose | 26 hours during closed-loop control
  No.
Continuous glucose monitored glycemic variability measured as SD | 26 hours during closed-loop control
  mmol/L
Continuous glucose monitored glycemic variability measured as CV | 26 hours during closed-loop control
  percentage
Composite outcome: Percentage of participants achieving (1) time in range (3.9-10) > 70 %, (2) time in alert hypoglycemia (<3.9 mmol/l) < 4 %, and (3) time in clinical hypoglycemia (<3.0 mmol) < 1% as measured by CGM and YSI | 26 hours during closed-loop control
  percentage
Total insulin dose | 26 hours during closed-loop control
  units
Total glucagon dose | 26 hours during closed-loop control
  mg
Number of manual insulin boluses | 26 hours during closed-loop control
  No.
Number of adverse events - Nausea | 26 hours during closed-loop control
  No of event if visual analog scale (0-100) increase >10 from baseline
Number of adverse events - Headache | 26 hours during closed-loop control
  No of event if visual analog scale (0-100) increase >10 from baseline
Number of adverse events - Palpitation | 26 hours during closed-loop control
  No of event if visual analog scale (0-100) increase >10 from baseline
Number of vomits | 26 hours during closed-loop control
  No of event if visual analog scale (0-100) increase >10 from baseline
Difference between actual and participant-estimated carbohydrate content in meals | 26 hours of closed-loop glucose control
  g per meal
Mean Borg scale | During 45 minutes exercise
  Scale of perceived exertion from 6 (no effort activity) to 20 (max effort activity)
Physical activity intensity measured by ActiGraph GT9X Link | 26 hours
  Percentage of sedentary activity
Sleep efficiency measured by ActiGraph GT9X Link | 26 hours
  The ratio of total sleep time to time in bed

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From 1 year to 10 years after completion

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT04949867/Prot_SAP_000.pdf